CLINICAL TRIAL: NCT06793397
Title: An Efficacy and Safety, Phase III, Multi-center, Double-Blind, Randomized Controlled Study Comparing 2 Active Doses of CYB003 and Placebo in Eligible Participants With Major Depressive Disorder
Brief Title: A Study of a Deuterated Psilocin Analog (CYB003) in Humans With Major Depressive Disorder
Acronym: EMBRACE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cybin IRL Limited (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYB003-003
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD); Depression in Adults; Depression - Major Depressive Disorder; Depression Disorders; Depression Disorder; Depression
Keywords: MDD; Psychedelic; Depression; Major Depressive Disorder; CYB003; CYB003-001; CYB003-002; Psilocybin; psilocin-7438
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental Arm A CYB003 in 2 of 2 Dosing Sessions (Experimental): Arm A participants will receive 8 mg of CYB003 in 2 of 2 medicine sessions, approximately three weeks apart. All Arm A participants will continue on their current antidepressants and receive psychological support throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychological Support
- Experimental Arm B CYB003 in 2 of 2 Dosing Sessions (Experimental): Experimental Arm B participants will receive 16 mg of CYB003 in 2 of 2 medicine sessions, approximately three weeks apart. All Arm B participants will continue on their current antidepressants and receive psychological support throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychological Support
- Placebo Comparator: Arm C Placebo in 2 of 2 Dosing Session (Placebo Comparator): Participants will receive placebo in 2 of 2 medicine sessions, approximately three weeks apart. All Arm C participants will continue on their current antidepressants and receive psychological support throughout the study. Non-responders will be eligible to receive CYB003 in a subsequent extension trial.
  Interventions: Behavioral: Psychological Support

INTERVENTIONS:
Drug: CYB003 — CYB003 is a deuterated psilocin analog.
  Arms: Experimental Arm A CYB003 in 2 of 2 Dosing Sessions; Experimental Arm B CYB003 in 2 of 2 Dosing Sessions
Behavioral: Psychological Support — Manualized psychological support performed by facilitator.

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability of CYB003 compared to matching placebo as adjunctive treatment in patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following criteria to be included in the trial:
* Age18 to 85 years.
* Participant has a diagnosis of MDD.
* Moderate to severe depression at Screening.
* Participants have been on a stable dose of antidepressant medication at an adequate dose in the last 4 weeks prior to Screening.
* Participant has a body mass index (BMI) of 40 kg/m2 or less (BMI ≤40 kg/m2), inclusive, at Screening.
* Participants with well controlled hypertension.
* Participant is able to refrain from smoking during the dosing session.
* Participants must use a condom plus spermicide during the trial and for 12 weeks afterwards.

Participants of childbearing potential must agree to use a highly effective method of and a negative pregnancy test at Screening and Day -1 prior to dosing.

* Participants of non-childbearing potential who are or were capable of producing eggs (ova) must have been postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.
* Participants have provided written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form.

Exclusion Criteria

* Participants with any of the following characteristics/conditions will be excluded from trial participation:
* Current or previously diagnosed schizophrenia spectrum or other psychotic disorders.
* Family history of schizophrenia, schizoaffective disorder, or bipolar disorder type 1 (first-degree relatives).
* Significant suicide risk within 12 months of Screening.
* Current or previous diagnosis of treatment-resistant MDD.
* Has had electroconvulsive treatment, transcranial magnetic stimulation, deep brain stimulation, or vagal nerve stimulation for any episode of MDD in the last 6 months.
* Currently receiving a monoamine oxidase inhibitor, tricyclic antidepressants, mirtazapine, trazodone, moclobemide, buspirone, or an antipsychotic or mood stabilizer.
* Clinically relevant history of abnormal physical health interfering with the trial (including but not limited to, neurological, cardiovascular, respiratory, gastrointestinal [including dyspepsia or gastroesophageal reflux disease], hepatic, or renal disorder).
* Has hypothyroidism or hyperthyroidism, unless controlled on appropriate medication.
* Current diagnosis of uncontrolled hypertension or an arrhythmia, or clinically relevant abnormal results for heart rate.
* Participants have a presence or relevant history of organic brain disorders.
* Participant is taking or has taken OTC doses of 5 hydroxytryptophan or St John's Wort within prior to trial medication administration.
* Strenuous exercise prior to each clinic visit.
* Donation of blood or plasma within 4 weeks prior to first dosing and until 4 weeks after final dosing.
* Participants capable of producing sperm who will not abstain from sperm donation between first dosing and 12 weeks after final dosing.
* Participants of childbearing potential who are pregnant, breastfeeding, planning to conceive or unwilling to abstain from egg (ova) donation between first dosing and 12 weeks after final dosing.
* History of serotonin syndrome.
* Unwilling to consent to audio and video recording of psychological support and dosing sessions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-03-18 (Estimated); Study Completion 2027-05-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Scale (MADRS) | Screening Day-45, Baseline, Day -1, Day 21, Day 42, Day 63 and Day 84/End of Trial.
  The MADRS is a 10-item scale with ratings based on a clinical interview which moves from broadly phased questions about symptoms to more detailed ones allowing a precise rating of severity.
  The total score ranges 0-60, higher scores denote greater severity.

SECONDARY OUTCOMES:
The Beck Depression Inventory - Second Edition (BDI-II) | Day -1, Day 21, Day 42 and Day 84/End of Trial.
  The Beck Depression Inventory-Second Edition (BDI-II) is a 21-question multiple-choice self-report inventory, assessing depressive symptoms and severity.
  Each question is scored on a scale value of 0 to 3, with higher total scores indicating more severe depressive symptoms. Each of the 21 items corresponding to a symptom of depression is summed to give a single score for the BDI-II, so the total score possible is 63 and minimum if everything is zero would be 0.
The Clinical Global Impression Scale (CGI-S) | Screening Day-45, Baseline Day -1, Day 42, Day 84/End of Trial.
  The Clinical Global Impression Scale is a clinician-rated instrument comprised of 3 global measures: severity of illness, global improvement and efficacy index.
  Only the severity of illness ang global improvement measures will be utilized for this trial.
  Higher score means more severe symptomology, worse outcome. CGI-S scoring is as follows:
  1. = Normal, not at all ill
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill patients
The Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline Day -1, Day 21, Day 42, Day 63 and Day 84/End of Trial.
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) is a 7-item self reported assessment that measures the severity of generalized anxiety disorder symptoms.
  Participants respond to each item using a 4-point scale from 0 to 3. Participants choose one of 4 severity scores associated with problems related to the common anxiety disorders to indicate the degree to which these problems caused functional and/or social difficulties. A total score is obtained by the sum of all total column values, higher scores indicate more functional/social impairment/difficulties. Score range is as follows:
  Scores represent:
  0 - 4 = Minimal anxiety 5 - 9 = Mild anxiety 10 - 14 = Moderately anxiety 15 - 21 = Severe anxiety
The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Day -1, Day 21, Day 42 and Day 84/End of Trial.
  The original Quality of Life Enjoyment and Satisfaction Questionnaire is a 93 item, participant facing, self reported measure used to evaluate intervention-related changes in quality of life, divided int the following sections: physical health, feelings, work, household duties, school, leisure time activities, social relations and general activities.
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) version will be used in this trial.
  Each item rated on a 5-point scale ranging from 1 (very poor) to 5 (very good), higher score indicates greater satisfaction. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70. So the minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mazer, Study Director — Cybin IRL Limited
Locations (67):
- United States (32):
  - UAB Psychiatry and Behavioral Neurology, Birmingham, Alabama
  - Lighthouse Psychiatry, Gilbert, Arizona
  - Pillar Clinical Research - Little Rock, Little Rock, Arkansas
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - CalNeuro Research Group, Los Angeles, California
  - ATP Clinical Research, Orange, California
  - NRC Research Institute, Orange, California
  - Inland Psychiatric Medical Group Inc (IPMG Research), San Juan Capistrano, California
  - Psychedelic Science Institute, Santa Monica, California
  - Stanford University, Stanford, California
  - Yale School of Medicine - Connecticut Mental Health Center (CMHC), New Haven, Connecticut
  - CNS Healthcare, Jacksonville, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Emory University Dept of Psychiatry and Behavioral Studies, Atlanta, Georgia
  - Psych Atlanta, Marietta, Georgia
  - Rush University, Chicago, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Institute for Integrative Therapies, Eden Prairie, Minnesota
  - Bio Behavioral Health, Toms River, New Jersey
  - New York State Psychiatric Institute, New York, New York
  - SP Research PLLC, Oklahoma City, Oklahoma
  - Adams Clinical Philadelphia, Philadelphia, Pennsylvania
  - Flourish Research Philadelphia, Philadelphia, Pennsylvania
  - Austin Clinical Trial Partners, Austin, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Brain Health Consultants and TMS Center, Houston, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Core Clinical Research, Everett, Washington
  - Seattle Neuropsychiatric Treatment Center, Seattle, Washington
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Thompson Brain & Mind Healthcare (TBMH), Maroochydore, Queensland
  - Ramsay Clinic, Melbourne, Victoria
  - Neurocentrix Research, Melbourne, Victoria
  - Monash University - Notting Hill, Notting Hill, Victoria
- Czechia (3):
  - Institute of neuropsychiatric Care (INEP), Prague
  - Psyon s.r.o., Prague
  - A-SHINE s.r.o., Předměstí
- Germany (4):
  - Universitätsklinikum des Saarlandes und Medizinische Fakultät der Universität des Saarlandes, Homburg, Saarland
  - Charité Universitaetsmedizin Berlin, Berlin
  - University Hospital Frankfurt, Frankfurt am Main
  - Central Institute of Mental Health, Mannheim
- Greece (3):
  - Eginitio Hospital, Athens
  - Attikon University Hospital, Athens
  - Papageorgiou General Hospital, Thessaloniki
- Ireland (2):
  - Sheaf House - Tallaght Adult Mental Health Service, Dublin
  - La Nua Day Hospital Mental Health Centre, Galway
- Poland (6):
  - Uniwersytecki Szpital Kliniczny W Białymstoku, Bialystok
  - Promente - Centrum Neurologii i Psychogeriatrii w Bydgoszczy, Bydgoszcz
  - UCK, Gdansk
  - Centrum Badan Klinicznych PI-House Sp. z o.o, Gdansk
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Department of Pharmacology and Physiology of CNS, Warsaw
- United Kingdom (12):
  - Cambridge University Hospital NHS, Cambridge
  - Clerkenwell Health - Doncaster, Doncaster
  - NHS Research Scotland, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - St Pancras Clinical Research, London
  - King's College London, London
  - Clerkenwell Health - Welbeck Street, London
  - Re:Cognition Health, London
  - Clerkenwell Health - Baker Street, London
  - Wolfson Unit - Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne
  - Ascend Clinical Research, Reading
  - Sheffield Health and Social Care NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Apply for Trial Here — http://embrace-mdd-trial.com/embracepublic/home/CT